CLINICAL TRIAL: NCT04753281
Title: Feasibility of a Multi Site RCT to Establish the Effectiveness of a Health Behaviour Change Intervention for Patients With Peripheral Arterial Disease (PAD).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 240417
Record Dates: First submitted 2021-02-03; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle counselling (Other): Participants will receive an assessment appointment and up to 8 follow up sessions with a Health Psychologist to help them set goals and monitor changes of their own self management behaviour.
  Interventions: Other: Lifestyle counselling
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Lifestyle counselling — brief psychological intervention, based on the behaviour change whee
  Arms: Lifestyle counselling

SUMMARY:
The purpose of this study was to evaluate the feasibility of conducting a randomised controlled trial (RCT) comparing brief psychological intervention to help patients with Peripheral Arterial Disease (PAD), reduce cardiovascular risk factors compared to control/treatment as usual in a vascular outpatient clinic. Trial feasibility was defined as the successful recruitment and retention of participants, adherence to the intervention, identification of barriers to the intervention and collection of clinical and quality of life outcome data. Qualitative data was collected to evaluate participant experience and the clinical impact of a supported self-management intervention delivered in a routine clinical setting.

DETAILED DESCRIPTION:
The aim of this study was to assess the feasibility of conducting a definitive multi-centre trial of a specially designed health behaviour change intervention delivered in a secondary care outpatient clinic to improve the primary clinical outcome of functional walking ability This feasibility study, based on the MRC framework for assessing feasibility and piloting methods, will assess the relative strengths and weaknesses of the intervention and study design, as well as pave the way for a larger and more definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Newly diagnosed with PAD resulting in claudication in one or both legs
* Reduced Ankle Brachial Index (ABI < 0.80).

Exclusion Criteria:

* Patients with an ABPI of less than 0.35, with rest pain or tissue loss were excluded and classified as cases of critical limb ischaemia requiring revascularisation.
* Severe mental health problems such as severe depression with suicidal ideation, psychosis, personality disorder
* Terminal illness
* Patients for whom it would be medically unadvisable to increase their daily walking (including heart failure, cancer, exercise induced asthma, unstable angina. Inability to walk unaided, history of orthopaedic surgery or significant bony disease impacting upon their mobility).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Functional walking ability | 1 year study
  To establish feasibility of a large scale RCT of a specifically designed health behaviour change intervention to improve functional walking ability in adults with PAD.
  We will use the standard measure of functional walking.

SECONDARY OUTCOMES:
Anxiety and Depression | 1 year
  The Chief Investigator (CI) will administer brief, self-report inventories at baseline, 3 months and 6 months follow-up to establish participants': anxiety and depression measured using Hospital Anxiety and Depression Scale, (HADS).
Emotional wellbeing | 1 year
  The Chief Investigator (CI) will administer brief, self-report inventories at baseline, 3 months and 6 months follow-up to establish participants': positive emotional wellbeing measured using the Warwick-Edinburgh Mental Wellbeing Scale Scored 1-5 (1 being none of the time and 5 being all of the time).
Health related quality of life | 1 year
  The Chief Investigator (CI) will administer brief, self-report inventories at baseline, 3 months and 6 months follow-up to establish participants': health-related quality of life measured using EQ-5D-5L *EQ-5D-5L Scored -10 -100. (-10 being the worst health you can imagine and 100 being the best health you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mccallum, Principal Investigator — NHSGRAMPIAM
Locations (1):
- NHS Grampian, Aberdeen, AB25 2ZP, United Kingdom

IPD SHARING:
Plan to Share IPD: No